CLINICAL TRIAL: NCT05669729
Title: A Survey Among Patients, Caregivers and Home Infusion Nurses Based in the European Union to Assess Their Awareness and Understanding of Educational Materials Supporting VPRIV® Infusion at Home
Brief Title: A Survey to Assess Participants', Caregivers', and Nurses' Use and Understanding of Educational Material on Velaglucerase Alfa (VPRIV) Home Infusion
Status: Not yet recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-669-4018
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Gaucher Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VPRIV® Home Infusion: Participants diagnosed with Gaucher disease will receive VPRIV® home infusion, administered by their caregivers and home infusion nurses will participate in the survey and complete the non-nominative web-based questionnaires on Day 1.

SUMMARY:
The main purpose of this survey is to determine participants', caregivers', and nurses' understanding and use of educational materials (EM) on VPRIV home treatment. EM includes an infusion diary and guide and an emergency plan related to VPRIV infusion given at home for Gaucher disease. The survey is conducted in European countries.

Data will be collected directly from participants, caregivers, and nurses in form of a questionnaire, electronic or paper.

DETAILED DESCRIPTION:
The participants diagnosed with Gaucher disease receiving VPRIV® home infusion, their caregivers and home infusion nurses were observed in this study. This cross-sectional study will determine and assess the understanding of the educational material (EM), including infusion diary and emergency plan associated with VPRIV® home infusion in participants diagnosed with Gaucher disease, their caregivers and home infusion nurses.

The study will recruit approximately 30 participants/caregivers and 30 home infusion nurses. The survey will be conducted through non-nominative web-based questionnaires that will be completed in approximately 10-15 minutes. All participants will be enrolled in a single observational group:

• VPRIV® Home Infusion

The trial will be conducted in home-based setting in Austria, Belgium, Finland, France, Germany, Italy, the Netherlands, and Spain.

ELIGIBILITY:
Inclusion criteria:

1. Gaucher disease participants who receive VPRIV® for home infusion and their caregivers.
2. Home infusion nurses administering VPRIV® to participants with Gaucher disease at home.

Exclusion criteria:

Potential respondents will be excluded if they have conflicts of interest with the survey (e.g., if they are employed by regulatory bodies, or pharmaceutical industry).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will recruit Gaucher disease participants receiving VPRIV® home infusion, their caregivers and home infusion nurses who administer VPRIV® infusion at home in European countries.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-09-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants and Caregivers Aware of Educational Material (EM) | Day 1
  EM includes home infusion guide, infusion diary, and safety and emergency plan.
Percentage of Participants and Caregivers who Understand the EM | Day 1
  EM includes home infusion guide, infusion diary, and safety and emergency plan.
Percentage of Participants and Caregivers who Utilize the EM | Day 1
  EM includes home infusion guide, infusion diary, and safety and emergency plan.
Percentage of Home Infusion Nurses Aware of the EM | Day 1
  EM includes home infusion guide, infusion diary, and safety and emergency plan.
Percentage of Home Infusion Nurses who Understand the EM | Day 1
  EM includes home infusion guide, infusion diary, and safety and emergency plan.
Percentage of Home Infusion Nurses who Utilize the EM | Day 1
  EM includes home infusion guide, infusion diary, and safety and emergency plan.

OTHER OUTCOMES:
Usefulness of the EM for Participants and Caregivers | Day 1
  EM includes home infusion guide, infusion diary, and safety and emergency plan. Usefulness will be assessed using the 12-item participant and caregiver questionnaire, and 15-item home infusion nurse questionnaire.
Usefulness of the EM for Home Infusion Nurses | Day 1
  EM includes home infusion guide, infusion diary, and safety and emergency plan. Usefulness will be assessed using the 12-item participant and caregiver questionnaire, and 15-item home infusion nurse questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/e895407fd93e49c7?idFilter=%5B%22TAK-669-4018%22%5D